CLINICAL TRIAL: NCT05767918
Title: StratosPHere: Optimal Biomarkers to Ascertain Target Engagement in Therapies Targeting the BMPR2 Pathway in Pulmonary Arterial Hypertension (PAH)
Brief Title: StratosPHere (Non-interventional Study)
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Medical Research Council (Other Government); University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: P02739
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Arterial Hypertension; Idiopathic Pulmonary Arterial Hypertension; Pulmonary Hypertension; Respiratory Disease
Keywords: Bone morphogenetic type 2 protein; BMPR2; Biomarker
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum and plasma samples - Peripheral blood mononuclear cells (PBMCs) were isolated from whole blood samples and the live cells cryogenically frozen pending analysis. Blood samples destined for RNA analysis were collected into Tempus Blood RNA tubes and stored at -80˚C pending RNA extraction and further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary Arterial Hypertension is a progressive disease that has no cure. Patients die young and are limited in their daily activity. Current treatments only treat the symptoms of the disease rather than the underlying cause. At least 1 in 5 patients has a change in a gene called the bone morphogenetic type 2 protein (or BMPR2). Extensive evidence supports the concept of addressing the reduced levels of the BMPR2 protein to reverse disease. Through work already undertaken by this group, two potential therapies which increase BMPR2 have been identified for use in a future randomised control trial. In order for a clinical trial to be informative we need an accurate way of measuring the protein or the effects of the protein (known as a biomarker). This study will use blood samples taken from 17 patients and 30 healthy participants over various time-points (2-5 visits over 5 weeks for healthy controls; 2 visits, approximately four months apart for patients). Laboratory work will help identify the best biomarkers for subsequent therapy studies. By defining the best biomarkers we can speed up the drug development in this rare disease.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a devastating and life-threatening disease that is associated with high morbidity and mortality. The disease is characterised by increased pulmonary arterial pressure; the blood pressure of the arteries found in the lungs. This increase in pressure is due to the progressive narrowing and obliteration of these blood vessels, often leading in failure of the right ventricle of the heart.

Current treatments for PAH utilise vasodilators to lessen the effects of the narrowing of the blood vessels and reduce blood pressure. However, a major breakthrough in our understanding of the molecular basis of PAH has been the identification of mutations, or changes, in important genes involved in the normal function of the lung vasculature. Mutations in the gene encoding bone morphogenetic protein type II receptor (BMPR2) have, to date been the most important genetic mutation identified, present in the majority (75%) of heritable PAH cases and approximately 11-44% of idiopathic cases (Dunmore et al). Such mutations result in a significantly reduced amount of this receptor on key cells in the pulmonary vasculature, the result of which is disruption of the normal cellular events and the subsequent development of vascular disease. Extensive research now exists on the role of BMPR2 in the development of PAH and pre-clinical findings support the targeting of BMPR2 as a potential treatment, however there are currently no therapeutics targeting the receptor in development.

To define the optimal biological biomarker end point of BMPR2 target engagement we will assess two study populations over a longitudinal time-course using peripheral blood samples.

Samples will be taken from a patient population with idiopathic or hereditary pulmonary arterial hypertension (n=17) and healthy volunteers (n=30) who will act as a control group.

Recruitment of healthy volunteers will be targeted at female aged 30-40 years as this is in line with the demographics of a typical PAH patient cohort. Blood samples will be collected from the control group across a total of 6 time points; the first 5 samples will be offered on a weekly basis with a final blood sample taken at 4 months. Sampling on weeks 2, 3, 4 and 16 will be optional. The expected duration for healthy volunteers is a total of 5 weeks with no follow up.

PAH participants will be sampled during routine clinic reviews over a four-month time period. Sampling will occur at separate two distinct time-points, three to six months apart. IPAH/HPAH participants will be recruited based upon their diagnosis and will be in WHO functional class I-IV and on stable medication or have unchanged PAH for at least one month prior to screening. The total duration for participants in this group will be approximately 3-6 months (typically 4 months), dependent on scheduling of clinical visits.

This will provide critical information for a future RCT testing two novel therapies with the potential to improve survival and quality of life for people diagnosed with PAH by providing a personalised approach to treatment.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* Individual must be 18 years of age or over
* Weigh > 40kg at screening visit / BMI under 35
* Healthy and well at each visit

PAH participants

* Must have a diagnosis of IPAH or HPAH with a WHO functional class I-IV
* Must be on stable or unchanged PAH therapeutics for at least one month prior to screening visit

Exclusion Criteria:

Health volunteers

* Known hepatitis B, HIV or tuberculosis
* Clinically severe anaemia or bleeding disorders

PAH participants

* Other forms of PH besides IPAH or HPAH
* Patients on TNF antagonists of other biological treatments
* Known hepatitis B, HIV or tuberculosis
* Clinically severe anaemia or bleeding disorders
* Female participants who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PAH patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Biomarker(s) identification | 2 years
  identify one or more biomarkers of increased BMPR2 expression or BMPR2 target engagement that fit a criterion of being reproducible and repeatable. We will define the acceptable level of variability of these in order to be used in the subsequent phase 2a trial that will be powered to detect a 30% increase in BMPR2, and or BMPR2 target engagement with an 80% power in the known patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Toshner Associate Professor MD FRCP, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge Heart and Lung Research Institute, Cambridge, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided